CLINICAL TRIAL: NCT05440656
Title: A Real World Multicenter 48 Week Prospective Cohort Study to Capture Clinical and Patient Centered Outcomes in Adults With Severe Eosinophilic Asthma Treated With Benralizumab in Routine Care Settings in Greece
Brief Title: A Real World Study to Capture Clinical and Patient Centered Outcomes in Adults With Severe Eosinophilic Asthma Treated With Benralizumab.
Acronym: EMPOWAIR
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3250R00102
Record Dates: First submitted 2022-06-13; First posted 2022-07-01 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Severe Eosinophilic Asthma
Keywords: Severe Asthma, Home Spirometry, Activity Tracker, Benralizumab
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: Cohort — Participants with Severe Eosinophilic Asthma

SUMMARY:
Severe eosinophilic asthma (SEA) is associated with poor disease control and compromised health-related quality of life (HRQoL), leading to a substantial psychosocial and economic disease burden. Benralizumab (Fasenra®), an interleukin (IL)-5-alpha receptor monoclonal antibody, is approved as an add-on maintenance treatment for SEA.

This study aims at collecting real-world data that extend beyond the clinical effectiveness of benralizumab to the participant-reported impact of treatment on their HRQoL, sleep quality, depression, anxiety, work productivity and activity impairment, but also on treatment effectiveness. Recent technological advances in portable spirometers and wearable activity trackers (WAT) to increase physical activity for participants with asthma, even for older participants, allow this study to collect data on lung function parameters and physical activity from such devices for the first time at a country level in Greece. Using a multi-aspect approach, this study will generate real-world evidence on a broad range of both well-established clinical and novel patient-centered outcomes which are critical to the assessment of the therapeutic benefit both from the physician's and the participant's perspective. All main study outcomes will be examined at various timepoints throughout the course of the 48-week observation period, starting as early as 4 weeks after treatment initiation, thus enabling the identification of 'early' treatment responders with a closer focus on patients' physical and psychological well-being and HRQoL in addition to asthma control and lung function metrics

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18 to 75 years (inclusive) at the time of benralizumab prescription
* Patients with physician-diagnosed Severe Eosinophilic Asthma SEA inadequately controlled despite high-dose inhaled corticosteroids (ICS) plus long-acting β-agonists (LABA)
* Patients who have been prescribed but not yet initiated treatment with benralizumab according to the Summary of Product Characteristics (SmPC), prior to signed Informed Consent, and for whom the decision to prescribe this therapy is clearly separated from the physician's decision to include the patient in the current study
* For patients that are not Oral Corticosteroid (OCS)-dependent: Blood eosinophil count (BEC) ≥150 cells/μL in the 2 weeks before benralizumab initiation and a historical value of ≥300 cells/μL during the previous year
* For OCS-dependent patients: BEC ≥150 cells/μL in the 2 weeks before benralizumab initiation or a historical value of ≥300 cells/μL during the previous year
* History of ≥1 documented Clinically Significant Exacerbations (CSE) in the 48 weeks prior to benralizumab initiation, and of ≥2 CSEs in the previous 24 months
* Patients must be willing and able to read and complete the study specific questionnaires
* Patients must be willing and able to use the study-specific wearable/handheld devices.

Note: This requirement applies only at the time of benralizumab (Fasenra®) prescription. If a patient stops using any or both of the aforementioned devices for any reason during his/her participation in the study, (s)he may continue participating in the study and this will not be considered as a reason for withdrawal.

-Patients must provide a written Informed Consent prior to inclusion to the study

Exclusion Criteria:

* Patients that meet any of the contraindications to the administration of the benralizumab outlined in the SmPC
* Concomitant treatment with any other biologic agent for any indication
* Previous exposure to anti-IL5/ILR5 treatment
* Exposure to omalizumab in the past 6 months prior to benralizumab initiation
* Clinically important pulmonary disease other than asthma or ever been diagnosed with any disease, other than asthma, that is associated with elevated BEC
* Acute upper or lower respiratory infections within 8 weeks prior to the date of informed consent
* Heavy smokers with a >20 pack-year smoking history
* Currently pregnant (or intention to become pregnant within the study period), breastfeeding or lactating women
* Known evidence of lack of adherence to asthma controller medications
* Use of immunosuppressive medication (including but not limited to: OCS [for reasons other than asthma], methotrexate, troleandomycin, cyclosporine, azathioprine, intramuscular long-acting depot corticosteroids [for reasons other than asthma] or any experimental anti-inflammatory therapy) within 3 months prior to the date of informed consent
* Patients who currently receive treatment with any investigational drug/device/intervention or who have received any investigational product within 30 days or 5 half-lives of the investigational agent (whichever is longer) before benralizumab initiation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Private practices and hospital clinics specializing in the management of asthma in geographically diverse locations throughout Greece
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-04-13 (Actual); Study Completion 2025-04-13 (Actual)

PRIMARY OUTCOMES:
Change in St. George's Respiratory Questionnaire (SGRQ) | 16 weeks after the initiation of the treatment
  Estimation of the proportion of patients achieving a minimum clinically important improvement in respiratory health status (≥ 4-point reduction from baseline in SGRQ total score) in SEA patients initiated on benralizumab

SECONDARY OUTCOMES:
Change in St. George's Respiratory Questionnaire (SGRQ) | 16 weeks after the initiation of the treatment
  Estimation of the proportion of patients achieving a moderately efficacious change in respiratory health status (≥ 8-point reduction from baseline in SGRQ total score)
Change in St. George's Respiratory Questionnaire (SGRQ) | after 4, 8, 32 and 48 weeks of treatment
  Estimation of the proportion of patients achieving a minimum clinically important improvement (≥ 4-point reduction in baseline SGRQ total score) and of those achieving a moderately efficacious change in respiratory health status (≥ 8-point reduction in baseline SGRQ total score)
Change in St. George's Respiratory Questionnaire (SGRQ) | after 4 and 48 weeks of treatment
  Determination of predictors of early clinically important improvement in respiratory health status (measured by the SGRQ) at 4 weeks of treatment with benralizumab, and at 48 weeks post-benralizumab initiation among the 4-week SGRQ responders
Change in ACQ-6 | after 4, 8, 16, 32, and 48 weeks of treatment
  Change in asthma control and the response rate as well as the response rate at 48 weeks post-benralizumab initiation among the 16-week ACQ-6 responders
Change in the annual rate of clinically significant exacerbations | between the 48-week periods pre- and post-benralizumab initiation
  Change in the annual rate of clinically significant exacerbations (CSE) and identification of factors influencing the CSE rate
change in asthma-related hospital-based health care resource utilization (HCRU) | between the 48-week periods pre- and post-benralizumab initiation
  Change in asthma-related hospital-based health care resource utilization (HCRU)
Change from baseline in clinic-measured spirometric lung function indices | after 16 and 48 weeks of benralizumab treatment
  Change from baseline in clinic-measured spirometric lung function indices and description of the FEV1 improvement rate at 48 weeks post-benralizumab initiation among patients who will achieve clinically meaningful improvement in FEV1 at 16 weeks post-benralizumab initiation
change from baseline in rescue medication use and in the proportion of nights with awakenings due to asthma requiring rescue medication use | after 4, 8, 16, 32 and 48 weeks of treatment
  Change from baseline in rescue medication use and in the proportion of nights with awakenings due to asthma requiring rescue medication use
change in cumulative oral corticosteroid (OCS) burden | etween the 16-week periods pre- and post-benralizumab initiation and the 48-week periods pre- and post-benralizumab initiation
  Change in cumulative oral corticosteroid (OCS) burden
change from baseline in anxiety and depression levels [assessed by the Hospital Anxiety and Depression Scale (HADS)] | after 16 and 48 weeks of treatment
  Change from baseline in anxiety and depression levels [assessed by the Hospital Anxiety and Depression Scale (HADS)]
change from baseline in patient-reported sleep quality [assessed by the Pittsburgh Sleep Quality Index (PSQI)] | after 16 and 48 weeks of treatment
  Change from baseline in patient-reported sleep quality [assessed by the Pittsburgh Sleep Quality Index (PSQI)]
change from baseline in work productivity and activity impairment [assessed by the Work Productivity and Activity Impairment:Respiratory Symptoms (WPAI:RS) questionnaire] | after 16 and 48 weeks of treatment
  Change from baseline in work productivity and activity impairment [assessed by the Work Productivity and Activity Impairment:Respiratory Symptoms (WPAI:RS) questionnaire]
clinician-assessed overall response to treatment using the Clinician Global Impression of Change (CGIC) | over the 48-week treatment period
  Clinician-assessed overall response to treatment using the Clinician Global Impression of Change (CGIC)
patient-perceived overall response to treatment using the Patient Global Impression of Change (PGIC) | after 48 weeks of treatment
  Patient-perceived overall response to treatment using the Patient Global Impression of Change (PGIC)
Percentage of patients remaining on treatment with benralizumab | at 48 weeks of treatment
  Treatment persistence rate on therapy
Percentage of patients having discontinued treatment with benralizumab | at 48 weeks of treatment
  Percentage of patients having discontinued treatment with benralizumab
description of reasons for treatment discontinuation | at 48 weeks of treatment
  description of reasons for treatment discontinuation
time to treatment discontinuation | at 48 weeks of treatment
  time to treatment discontinuation

CONTACTS AND LOCATIONS:
Locations (7):
- Greece (7):
  - Research Site, Alexandroupoli
  - Research Site, Athens
  - Research Site, Corfu
  - Research Site, Heraklion
  - Research Site, Ioannina
  - Research Site, Rio
  - Research Site, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home